CLINICAL TRIAL: NCT03716063
Title: Evaluation and Mechanism of Strengthening the Spleen and Reducing Phlegm Method in Improving Radical Resection Rate of Colorectal Cancer
Brief Title: Strengthening the Spleen and Reducing Phlegm Method in Improving Radical Resection Rate of Colorectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Chinese Academy of Medical Sciences (Other); Tianjin People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: httxixi
Record Dates: First submitted 2018-10-08; First posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; traditional Chinese medicine
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This study was double-blind. According to the randomized results, the experimental group was given orally therapeutic granules, while the control group was given orally low-dose granules.
Who Masked: Participant, Care Provider
Masking Description: This study was double-blind. According to the randomized results, the experimental group was given orally therapeutic granules, while the control group was given orally low-dose granules. Random sequence was generated by professional statisticians of group leader unit by statistical software. 350 subjects were divided into experimental group and control group according to the ratio of 1:1, 175 cases in each group. Random seeds and random sequences are stored as confidential data in opaque envelopes, and emergency envelopes are handed over to a third party to ensure that patients, researchers and outcome evaluators are unaware of the patient group before blindness is uncovered. After successful screening and signing the informed consent form, the patient can open a random envelope in turn and record the subject's name, hospital number and admission time on the envelope.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): The test group will oral Jianpi Huatan dispensing granule , once a day in the morning and evening, once a month for a course of treatment, a total of three courses.
  Interventions: Drug: Jianpi Huatan dispensing granule
- control group (Placebo Comparator): The control group will oral drug:low-dose control granules (containing 1/10 of the dose of the experimental group) , once a day in the morning and evening, once a month for a course of treatment, a total of three courses
  Interventions: Drug: Jianpi Huatan dispensing granule

INTERVENTIONS:
Drug: Jianpi Huatan dispensing granule — once a day in the morning and evening, every month for a course of treatment, a total of three courses

SUMMARY:
This study will take disease-free survival time and recurrence and metastasis rate as the main evaluation indexes, to evaluate the clinical efficacy of strengthening the spleen and reducing phlegm method in patients with stage II high-risk and stage III colorectal cancer

DETAILED DESCRIPTION:
The study enrolled 350 patients with stage II high-risk and stage III colorectal cancer who underwent adjuvant chemotherapy (based on a 5-fluorouracil（5-FU） regimen for at least 3 months) and patients who received chemotherapy for less than 3 months. The study will use a large sample, multicenter, randomized, double-blind study. The experimental group was given oral Jianpi Huatan dispensing granule, once a day in the morning and evening, 1 course per 1 month, a total of 3 courses; the control group of oral Chinese medicine formula low dose control granules (including the test group dose 1 /10), 1 time each morning and evening, 1 course per month, for a total of 3 courses.

The patients were followed up once a month during the treatment period and once every 3-6 months after the end of treatment until the patient relapsed, died or the study was over.Some patients in the study will be tested for circulating tumor cells.

Main outcome measures is Disease-free survival time（DFS）and Metastasis recurrence rate in 1 year；Secondary outcome measures：Quality of life score: applied quality of life scale.Metastasis recurrence rate in 2、3years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with colorectal cancer with clear pathological diagnosis and Western medicine diagnostic criteria；
2. Radical resection of colorectal cancer was performed and adjuvant chemotherapy (based on 5-FU regimens for at least 3 months) was completed within 3 months of the end of chemotherapy；
3. Tumor Node Metastasis(TNM) stage is high-risk II stage and III stage；
4. Age 18-80 years, sex unlimited；
5. No recurrence or metastasis by imaging or doctor's clinical judgement；
6. Signed informed consent； Note * According to National Comprehensive Cancer Network(NCCN )clinical guidelines: Phase II:T3-4N0M0; High-risk Phase II is defined as follows:：a.T4;b. Less than 12 lymph nodes were detected；c. preoperative intestinal obstruction, perforation of tumor site；d. poor histological differentiation (except highly unstable microsatellite)；e. neurological invasion and vascular tumor thrombus； f. positive or unknown margin, and insufficient margin safety distance. Phase III：T1-4N1-2M0.

Exclusion criteria:

1. History of previous or combined malignancies except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix；
2. Combined with severe heart, liver and kidney disease；
3. Any unstable condition or condition that may endanger patient safety and compliance with research, such as pregnancy, depression, manic-depressive disorder, obsessive-compulsive disorder, or schizophrenia;
4. The researchers determine that they were not suitable for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2018-10-30 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival time | 3 years
  from the date of radical resection of colorectal cancer to the time of recurrence or metastasis.
Metastasis recurrence rate in 1 year | 1 year
  The ratio of metastasis and recurrence to the patients was observed.

SECONDARY OUTCOMES:
Traditional Chinese Medicine(TCM )symptom grading table | 3 months
  Effective: after treatment, TCM symptom score decreased by more than 50% compared with that before treatment.
  Effective: decrease < 50% and equal to 30%; Invalid: decrease < 30%. Note: the formula is: (before treatment - integral after treatment) / before treatment by 100%
Functional Assessment of Cancer Therapy-Colorectal (FACT-C) scale | 3 months
  The FACT-C scale was divided into five grades: none (0), one point (1), some (2), equivalent (3) and very (4). The positive items (i.e. the higher the grade, the better the quality of life.)
Edmonton Symptom Assessment Scale( ESAS ) | 3months
  The scale used digital scoring method, each symptom scoring range of 0-10 points, 0 points for asymptomatic, 10 points for the most serious degree imaginable, patients choose a number to express their subjective feelings, the larger the number indicates the more serious the symptoms. 1~10 points were divided into 3 degrees, mild, moderate and severe. 1~3 were mild, 4~6 were moderate, and 7~10 were severe
Metastasis recurrence rate in 2 years | 2 years
  The ratio of metastasis and recurrence to the patients was observed.
Metastasis recurrence rate in 3 years | 3 years
  The ratio of metastasis and recurrence to the patients was observed.

CONTACTS AND LOCATIONS:
Overall Officials: yufei yang, doctor, Study Chair — Xiyuan Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Xiyuan Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li L, Qu Q, Cui N, Cai L, Zou J, Wu J, Hao T, Wu Y. Efficacy of jianpi huatan granule in reducing colorectal cancer metastasis and recurrence after radical resection and adjuvant chemotherapy: Study protocol for a randomised, double-blind, placebo-controlled, multicentre trial. Front Pharmacol. 2022 Sep 13;13:944475. doi: 10.3389/fphar.2022.944475. eCollection 2022. PMID 36176445